CLINICAL TRIAL: NCT05710497
Title: Assessing the Correlation of Maxillary Vascular Canal Thickness With Intraoperative Bleeding During Open Sinus Floor Augmentation: A Volumetric Tomography Study.
Brief Title: Maxillary Vascular Canal Thickness and Sinus Augmentation Bleeding
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ferit Bayram, Assist. Prof., Marmara University
Other Study IDs: MUDHF_FB_004
Record Dates: First submitted 2023-01-25; First posted 2023-02-02 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Bone Loss
Keywords: Maxillary Sinus Floor Augmentation; Volumetric Computed Tomography; Intra-operative bleeding
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the relationship between the maxillary intra-osseous vascular canal thickness as measured by volumetric tomography and the amount of intra-operative bleeding during open sinus floor augmentation. A sample of patients will be selected, and their maxillary intra-osseous vascular canal thickness will be measured using volumetric tomography. Intraoperative bleeding will be recorded during open sinus floor augmentation. The data will be analyzed to determine if there is a correlation between the thickness of the maxillary intra-osseous vascular canal and intraoperative bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Maxillary partial or total edentulism, including premolar/molar regions
* Medically healthy
* 2 to 5 mm residual bone height
* Sufficient bone width to place a standard dental implant (diameter >4mm)
* Age: 18-65 years
* Patients who volunteered to participate in the study and signed written informed consent

Exclusion Criteria:

* Maxillary sinusitis
* Acute myocardial infarction in the last 12 months
* Use of any medication that may inhibit bone healing
* History of radiotherapy in the head and neck region
* Presence of psychiatric problems
* Smoking more than 10 cigarettes a day
* Alcoholism
* Chronic drug use

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who present with the complaint of tooth loss in the posterior region and need rehabilitation with fixed prostheses on implants, whose horizontal bone width is suitable for dental implant placement but sinus floor augmentation will be performed due to insufficient vertical height.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Total amount of intraoperative bleeding | From beginning of surgery to end of surgery
  After surgery, the total amount of intraoperative bleeding will be calculated in milliliters.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chanavaz M. Sinus grafting related to implantology. Statistical analysis of 15 years of surgical experience (1979-1994). J Oral Implantol. 1996;22(2):119-30. PMID 9151634
- [Background] Elian N, Wallace S, Cho SC, Jalbout ZN, Froum S. Distribution of the maxillary artery as it relates to sinus floor augmentation. Int J Oral Maxillofac Implants. 2005 Sep-Oct;20(5):784-7. PMID 16274154
- [Background] Mardinger O, Abba M, Hirshberg A, Schwartz-Arad D. Prevalence, diameter and course of the maxillary intraosseous vascular canal with relation to sinus augmentation procedure: a radiographic study. Int J Oral Maxillofac Surg. 2007 Aug;36(8):735-8. doi: 10.1016/j.ijom.2007.05.005. Epub 2007 Jul 12. PMID 17629462
- [Background] Rosano G, Taschieri S, Gaudy JF, Del Fabbro M. Maxillary sinus vascularization: a cadaveric study. J Craniofac Surg. 2009 May;20(3):940-3. doi: 10.1097/SCS.0b013e3181a2d77f. PMID 19461336
- [Background] Rosano G, Taschieri S, Gaudy JF, Weinstein T, Del Fabbro M. Maxillary sinus vascular anatomy and its relation to sinus lift surgery. Clin Oral Implants Res. 2011 Jul;22(7):711-715. doi: 10.1111/j.1600-0501.2010.02045.x. Epub 2010 Dec 9. PMID 21143535
- [Background] Solar P, Geyerhofer U, Traxler H, Windisch A, Ulm C, Watzek G. Blood supply to the maxillary sinus relevant to sinus floor elevation procedures. Clin Oral Implants Res. 1999 Feb;10(1):34-44. doi: 10.1034/j.1600-0501.1999.100105.x. PMID 10196788
- [Background] Stern A, Green J. Sinus lift procedures: an overview of current techniques. Dent Clin North Am. 2012 Jan;56(1):219-33, x. doi: 10.1016/j.cden.2011.09.003. PMID 22117952
- [Background] Tatum H Jr. Maxillary and sinus implant reconstructions. Dent Clin North Am. 1986 Apr;30(2):207-29. PMID 3516738
- [Background] Zijderveld SA, van den Bergh JP, Schulten EA, ten Bruggenkate CM. Anatomical and surgical findings and complications in 100 consecutive maxillary sinus floor elevation procedures. J Oral Maxillofac Surg. 2008 Jul;66(7):1426-38. doi: 10.1016/j.joms.2008.01.027. PMID 18571027